CLINICAL TRIAL: NCT06196333
Title: Evaluation of Corneal Endothelium by Specular Microscope in Elderly Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Hennis Mahrous, Resident doctor, Assiut University
Other Study IDs: 04-2023-200228
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Evaluation of Corneal Endothelium in Elderly Diabetic Patient

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Diabetes: Diabetes patients above 40 years
  Interventions: Device: Non-contact specular microscopy
- Controls: Healthy controlled human beings have no medical histories
  Interventions: Device: Non-contact specular microscopy

INTERVENTIONS:
Device: Non-contact specular microscopy — using specular microscope to do morphological examination of corneal endothelial cells

SUMMARY:
A low endothelial count with endothelial pump dysfunction can contribute to corneal stromal hydration and loss of vision that can only be reversed by corneal transplantation,so this research proposed to detect any corneal endothelial changes related to DM , its duration and control of diabetes.

DETAILED DESCRIPTION:
- To establish any correlation between endothelial changes , and the duration of diabetes, hemoglobin A1c (HbA1c) by using specular microscope to do morphological examination of corneal endothelial cells, makes the measurement of mean cell density (MCD), measurement of coefficient of variation (CV) in the cell size as well as hexagonal appearance of the cell. These parameters provide the functional status index of the corneal endothelial layer .

ELIGIBILITY:
Inclusion Criteria:

* - Diabetic patient type 2
* Elderly patients above 40 years old

Exclusion Criteria:

* - Patients with any of the following conditions have been omitted from the study included a past medical history of ocular trauma, corneal or intraocular inflammation, the use of systemic drugs that could affect endothelial cells, evidence of endothelial disease during a slit-lamp examination, previous ocular surgery (including cataract surgery), increased intraocular pressure, corneal opacity, or retinal photocoagulation procedures.
* non of the inclusion criteria patients

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Not gender based from 40 years to 80 years diabetic patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2024-11-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Endothelial count | 15 months
  Corneal endothelial cell count, coefficient of variation, percentage of hexagonal cells and central corneal thickness will be evaluated and correlated to known normal values in the same healthy individual age group

SECONDARY OUTCOMES:
Correlated change | 15 months
  Correlated change of corneal endotheliam to duration and control of DM